CLINICAL TRIAL: NCT00004922
Title: A Phase II Clinical Trial of Irinotecan (CPT-11) in Patients With Advanced High Grade Neuroendocrine Tumors
Brief Title: Irinotecan in Treating Patients With Advanced Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-041; CDR0000067605 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1683
Record Dates: First submitted 2000-03-07; First posted 2003-10-01 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Carcinoma of Unknown Primary; Neuroendocrine Carcinoma; Neuroendocrine Carcinoma of the Skin
Keywords: newly diagnosed carcinoma of unknown primary; recurrent carcinoma of unknown primary; stage III neuroendocrine carcinoma of the skin; recurrent neuroendocrine carcinoma of the skin; neuroendocrine carcinoma
MeSH Terms: conditions — Neoplasms, Unknown Primary; Carcinoma, Neuroendocrine; Carcinoma, Merkel Cell | interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have advanced neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of irinotecan in terms of tumor response, time to tumor progression, and survival in patients with advanced high grade neuroendocrine tumors.
* Evaluate the dose limiting and nondose limiting toxicities of this treatment regimen in this patient population.

OUTLINE: Patients receive irinotecan IV over 90 minutes once weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed until death.

PROJECTED ACCRUAL: A total of 10-31 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic or unresectable high grade neuroendocrine tumor including:

  * Small cell carcinoma
  * Large cell neuroendocrine carcinoma
  * Other high grade neuroendocrine carcinomas without specification to cell size
  * No lung only involvement without any other primary site
* No primary small cell lung cancer with or without metastases
* Bidimensionally measurable disease with at least one lesion measuring at least 1 cm by 1 cm
* High grade tumor indicated by at least one of the following:

  * Growth pattern suggestive of neuroendocrine differentiation
  * Mitotic rate greater than 15 mitoses per 10 hpf
  * Presence of abundant necrosis
* Immunohistochemical evidence of neuroendocrine differentiation by positive staining for chromogranin, synaptophysin, or neuron specific enolase if no classic microscopic appearance of small cell carcinoma
* No low grade neuroendocrine tumors (e.g., carcinoid tumors, pancreatic endocrine tumors) and atypical tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT no greater than 5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No uncontrolled congestive heart failure requiring therapy

Other:

* No active or uncontrolled infection
* HIV negative
* No psychiatric or other disorder that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 2 prior chemotherapy regimens
* No prior camptothecins

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States